CLINICAL TRIAL: NCT04614896
Title: Use of Transoral Ultrasound for Measuring Depth Of Invasion in Oral Tongue Carcinoma, and Comparing Obtained Measurements With Measurements From MRI With the Results Obtained From Pathological Examination of Surgically Resected Specimens
Brief Title: Use of Ultrasound for Measuring Size of Oral Tongue Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mikkel Kaltoft, Consultant, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Ultrasoundfortonguetumors
Record Dates: First submitted 2020-10-28; First posted 2020-11-04 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Tongue SCC; Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound for measuring DOI in tongue tumors (Experimental): All patients included with tongue carcinoma
  Interventions: Diagnostic Test: Transoral ultrasound of tongue tumors

INTERVENTIONS:
Diagnostic Test: Transoral ultrasound of tongue tumors — A transoral ultrasound scan of tongue tumors will be performed to assess the depth of invasion of the tumor

SUMMARY:
The purpose of this study is to investigate the use intraoral ultrasound for measuring depth of invasion (DOI) in oral tongue squamous cell carcinoma. The DOI's measured on ultrasound and measurements from MRI scans, will be compared to the measurements made from pathological examination of removed specimens.

DETAILED DESCRIPTION:
The investigators will conduct a prospective cohort study to investigate the correlation between DOI measurements from preoperative imaging (MRI and intraoral ultrasound), and final histopathology findings.

All patients with oral tongue cancer histologically verified on biopsy diagnosed in the Capital Region and Zealand Region (population 2.6 mio) are treated at the department of Head and Neck surgery at Copenhagen University Hospital (Rigshospitalet). These patients will be invited to participate in the study before or at their multidisciplinary team (MDT) conference at Rigshospitalet where the final treatment will be decided.

The ultrasound exam is conducted with a bk5000 or bk3000 machine, a "Hockey Stick" X18L5s transducer or a 18L5s Linear transducer.

The transducer will be placed directly on the tongue tumor. The tumor size will be measured, and depth of invasion will be estimated. For later reevaluation of the ultrasound images, a sweep will be performed, and image files and video clips will be stored for documentation.

Patients will primarily be examined in the outpatient clinic, and the measurement will be repeated at the time of surgery when the patient is in general anesthesia. It is, however, at time of the examination outpatient clinic that the information about DOI is most useful in planning the treatment, and therefore this is measurement the investigators will be focusing on.

Each MRI scan will be reviewed by a radiologist and the DOI will be assessed if possible. According to the AJCC Cancer Staging System, 8th edition, "DOI is measured by first finding the 'horizon' of the basement membrane of the adjacent squamous mucosa. A perpendicular 'plumb line' is established from this horizon to the deepest point of tumor invasion" [AJCC ]

The investigators aim to include 30 Patients in this study. The annual number of patients in our clinic operated for oral tongue carcinoma is around 50, so the investigators aim to include the 30 patients within one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with squamous cell carcinoma on the lateral tongue

Exclusion Criteria:

* Patients with tumor elsewhere in the oral cavity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Correlation of DOI measured on ultrasound and on MRI compared to pathological examination | when pathological examination is made, within 4 weeks of US and MRi
  Measurement of DOI in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Kaltoft, MD, Principal Investigator — Consultant
Locations (1):
- Rigshospitalet Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No